CLINICAL TRIAL: NCT02844829
Title: Improved Prostate Cancer Diagnosis - Combination of Rapid Prebiopsy Magnetic Resonance Imaging and Biomarkers
Acronym: IMPROD2_0
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Hannu Aronen, Professor, Chief Physician, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: T166/2016
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Magnetic Resonance Imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI and biomarkers (Other): Prostate MRI. Blood and urine biomarkers. Both prior to biopsy. Tissue samples during prostatectomy.
  Interventions: Other: Prostate MRI

INTERVENTIONS:
Other: Prostate MRI — MRI of the prostate prior to prostate biobsy

SUMMARY:
This study will enroll 200 men with clinical suspicion of prostate cancer due to higher serum level of PSA than 2.5 ng/ml or abnormal digital rectal examination.

Anatomical magnetic resonance imaging (MRI) and diffusion weighted imaging (DWI) at 3 Tesla (T) magnetic field using surface coils will be used to non-invasively predict the presence or absence of prostate cancer.

Targeted TRUS guided biopsy based on MRI findings will be performed in addition to routine twelve core TRUS biopsy.

Moreover, selected serum and urine biomarkers as well as biomarkers extracted from fresh biopsy sample will be collected and correlated with the presence or absence of prostate cancer.

DETAILED DESCRIPTION:
Specific aims of the current study are as follows:

i) To determine the sensitivity, specificity and accuracy of a novel rapid anatomical MRI and DWI at 3T magnetic field for the detection of prostate cancer in correlation with systematic TRUS guided biopsy

ii) To determine the sensitivity, specificity and accuracy of selected serum, urine and tissue biomarkers for detection of prostate cancer

iii) To develop statistical model for diagnosis of prostate cancer incorporating findings of a novel rapid MRI/DWI and selected biomarkers

iv) To assess the applicability of TRUS guided prostate biopsy based on MRI finding in patient with no previous prostate biopsy

v) To develop and validate an imaging protocol which will become the standard protocol for prostate imaging at Medical Imaging Centre of Southwest Finland (VSKK) / TYKS, Turku, Finland.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40 to 85 years
* Language spoken: Finnish
* Clinical suspicion of prostate cancer, based on: serum level of PSA from 2,5 ng/ml to 25 ng/ml in two following measurements and/or abnormal digital rectal examination
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethics Committee (EC) approved informed consent documents in the presence of the designated staff

Exclusion Criteria:

* previous prostate biopsies
* previous diagnosis of prostate carcinoma
* previous prostate surgeries, e.g. TURP (transurethral prostatic resection)
* symptomatic of acute prostatitis
* contraindications for MRI (cardiac pacemaker, intracranial clips etc)
* uncontrolled serious infection
* claustrophobia
* any other conditions that might compromise patients safety, based on the clinical judgment of the responsible urologist

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity and accuracy of MRI and DWI at 3T magnetic field for the detection of prostate cancer in correlation with systematic TRUS guided biopsy | Baseline (MRI prior to prostate biopsy)

SECONDARY OUTCOMES:
Sensitivity, specificity and accuracy of selected serum, urine and tissue biomarkers for detection of prostate cancer | Baseline and during procedure
  Serum and urine samples before prostate biopsy and tissue samples during prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Hannu J Aronen, M.D. Ph.D., Principal Investigator — Diagnostic radiology University of Turku
Locations (1):
- Department of Urology, Turku University Hospital, Turku, Western Finland Province, Finland

IPD SHARING:
Plan to Share IPD: Undecided